CLINICAL TRIAL: NCT05694832
Title: Assessing the Impact of Expressive Writing as a Nonpharmacologic Therapeutic Intervention Within a New Support Group for Patients With Cutaneous Graft-versus-Host Disease (EXPRESS-C-GVHD): A Pilot Trial
Brief Title: Expressive Writing in GVHD
Acronym: EXPRESS-C-GVHD
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jennifer Nam Choi, MD, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 21H12
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Expressive writing weekly session (Experimental): Weekly, 1-hour sessions of creative writing, discussion and social support, in a group setting via videoconference for a total of 4 sessions.
  Interventions: Behavioral: Expressive Writing

INTERVENTIONS:
Behavioral: Expressive Writing — Creative writing, discussion and social support, in a group setting via videoconference

SUMMARY:
Graft-versus-host-disease (GVHD) is a disease phenomenon that occurs when immune cells of the donor recognize and attack healthy tissue within the transplant recipient, or host. It is ultimately the result of the same immunological mechanisms that provide benefit to patients receiving hematopoietic stem cell transplantation (HSCT). In patients with hematologic malignancies, HSCT can be therapeutic, as donor T cells recognize and mount a response against cancerous cells. HSCT is also used in the setting of certain immunodeficiencies and inborn errors of metabolism for which therapeutic benefit is found in immunologic repletion.

To our knowledge, support groups have yet to be investigated in academic literature as a nonpharmacologic, therapeutic intervention for cutaneous GVHD patients to improve their distress, systemic disease, and quality of life. Given the dearth of research on nonpharmacologic therapies for cutaneous GVHD that address quality of life impairments, we seek to characterize the effect of an expressive writing and peer helping intervention contextualized within the framework of a support group. The primary goal of this study is to provide preliminary efficacy data of expressive writing as an intervention in patients with cutaneous GVHD to trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an active or previously diagnosed chronic cutaneous graft-versus-host disease (cGVHD).
* Patients must be age ≥18 years.
* Patients must be able to write using a utensil and paper or be able to type.
* Patients must have access to internet or cellular connectivity with sufficient bandwidth to participate in videoconferences (Zoom).
* Patients should be able to and planning to attend all four live videoconferencing sessions for the support group via Zoom.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with limited level of oral and written English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-01-21 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Change in Dermatology Life Quality Index scores | 4 weeks
  Measured at baseline and post completion of the 4 week expressive writing sessions

SECONDARY OUTCOMES:
Change in Short Form-36 scores | 4 weeks
  Measured at baseline and post completion of the 4 week expressive writing sessions

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Choi, Principal Investigator — Northwestern University
Locations (1):
- Department of Dermatology, Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaundinya T, Kye Y, El-Behaedi SE, Choi JN. Protocol for a feasibility trial (EXPRESS-C-GVHD) for an expressive helping intervention within a support group for cutaneous graft-versus-host-disease. Arch Dermatol Res. 2023 Dec;315(10):2905-2912. doi: 10.1007/s00403-023-02718-y. Epub 2023 Sep 12. PMID 37698591